CLINICAL TRIAL: NCT02891018
Title: A Multicenter, Prospective and Randomized Controlled Clinical Study (VasoguardTM Trial II) That Comparing the Safety and Efficacy of Paclitaxel Controlled Release Balloon Catheter (VasoguardTM) in the Treatment of In-stent Restenosis of Coronary Artery Lesion With Paclitaxel Release Coronary Balloon Catheter (SeQuent Please)
Brief Title: Comparing the Safety and Efficacy of Paclitaxel Controlled Release Balloon Catheter in the Treatment of In-stent Restenosis of Coronary Artery Lesion With Paclitaxel Release Coronary Balloon Catheter
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Branden-123456
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: In-stent Restenosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- paclitaxel controlled release balloon catheter (Experimental): Patients treated with paclitaxel controlled release balloon catheter
  Interventions: Device: paclitaxel controlled release balloon catheter Vasoguard TM
- paclitaxel release coronary balloon catheter (Experimental): Patients treated with paclitaxel release coronary balloon catheter
  Interventions: Device: paclitaxel release coronary balloon catheter SeQuent Please

INTERVENTIONS:
Device: paclitaxel controlled release balloon catheter Vasoguard TM
  Arms: paclitaxel controlled release balloon catheter
Device: paclitaxel release coronary balloon catheter SeQuent Please
  Arms: paclitaxel release coronary balloon catheter

SUMMARY:
Study purpose The safety and efficacy of paclitaxel controlled release balloon catheter Vasoguard TM in treatment of in-stent restenosis.

Study group Experimental group: paclitaxel controlled release balloon catheter Vasoguard TM Control group: paclitaxel release coronary balloon catheter SeQuent Please

ELIGIBILITY:
Inclusion Criteria:

- Subject need 18 to 80 years of aged male or non-pregnant women; Subject has stable anina pectoris, or unstable anina pectoris, or old myocardial infarction patients, or ischemia with evidence but without symptom; Subject has a life expectancy of more than 2 years; Subject occurred restenosis after vessel lesion in situ receiving the first stent operation; In-stent restenosis type Mehran I, II, III, IV, reference vessel diameter of 1.5-4.0 mm, length of 40 mm or less; Target lesion stenosis must be equal or greater than 70% or 50% and with evidence of ischemia; Single or two coronary small vessel lesions in situ; Other lesion which need interventional treatment must be away from target lesion at least 10 mm; Subject can understand the trail purpose, sign informed consent voluntarily, agree to accept clinical telephone follow-up and angiographic follow-up at 9 months; Target lesion can be pre-expanded successfully (Guide wire can get through lesion, balloon pre-expand the remnant stenosis of vessel lumen is less or equal to 50%, without current limiting interlayer and thrombosis).

Exclusion Criteria:

- Patient that in the opinion of the investigator is not appropriate for this trail; Pregnancy and lactation female patients; Patient has a life expectancy of less than 2 years; Severe congestive heart failure or NYHA IV heart failure; Patient who have bleeding constitution, cannot use anticoagulation and antiplatelet drugs; Patient that happened acute myocardial infarction within a week; Patient who happened stroke within six months; Patient who with severe renal failure (GFR≤30ml/min); Patient who had received heart transplantation; Patient who cannot tolerate aspirin and / or P2Y12 receptor inhibitor drugs; Patient who has allergy to paclitaxel, PLGA or contrast agent; Peptic ulcer or gastrointestinal bleeding within the prior 6 months. Patients who are participating in another drug or device clinical trail, which have not completed the primary endpoint follow- up period.

Angiographic relevant： Three or more coronary artery vessel lesion; Target vessel has extensive thrombosis evidence; Restenosis of vein graft after bypass surgery; Left main coronary artery and ostial lesion within 2mm; Target lesion proximal exist seriously distorted or severe calcified lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss | at 9 months

SECONDARY OUTCOMES:
Device Success Rate | at 9 months
Operation Success Rate | at 9 months
Target lesion in-segment rate after operation 9 months | at 9 months
Target lesion revascularization (TLR) and Target vessel revascularization (TVR) by clinical-driven | at 9 months
Major adverse cardiovascular events (MACE) related with device, include cardiac death, myocardial infarction of target vessel and target lesion revascularization (TLR) by clinical-driven | at 9 months
Thrombotic events incidence (ARC definition include deterministic thrombosis, possible thrombosis and not eliminating thrombosis; point-in-time include acute within 24h, subacute between 2 and 30 d and later period over 30 d) | at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Beijing, Beijing Municipality, China